CLINICAL TRIAL: NCT03470272
Title: Effects of Red Light LED Therapy on Body Contouring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Manamed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Manamed
Record Dates: First submitted 2017-12-14; First posted 2018-03-19 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active Device (Experimental): Active Device: The FB Professional LED red light therapy system
  FB Professional is a treatment regime using the FB Professional device for fat removal using red light therapy.
  Intervention device: FB Professional LED red light therapy is a non-invasive dermatological aesthetic treatment for the reduction of circumference of hips, waist and thighs.
  Interventions: Device: FB Professional LED Red light therapy; Device: Effects of Red Light LED Therapy on Body Contouring

INTERVENTIONS:
Device: FB Professional LED Red light therapy — FB Professional LED red light therapy is a non-invasive dermatological aesthetic treatment for the reduction of circumference of hips, waist and thighs. Measure before and after effects of device unit. Three measurements before of circumference of abdomen area and three measurements after comparing the results.
  Other Names: Effects of Red Light LED Therapy on Body Contouring
Device: Effects of Red Light LED Therapy on Body Contouring — Intervention is to take a sample and measure before and after using a sham unit (placebo) and take three measurements of abdominal before treatment and three measurements after sham treatment and compare to controlled treatment.

SUMMARY:
Red light laser therapy using 635nm red light laser technology has previously been shown to cause lipolysis in subcutaneous fat as a non-surgical method to promote weight loss and body contouring. This study hypothesizes that red LED light therapy using 650nm red light LED (light emitting diode) technology produces similar results to the laser device (red LASER 635nm) when preformed using a specified treatment protocol.

DETAILED DESCRIPTION:
Red light laser therapy using 635nm red light laser technology has previously been shown to cause lipolysis in subcutaneous fat as a non-surgical method to promote weight loss and body contouring. This study hypothesizes that red LED light therapy using 650nm red light LED (light emitting diode) technology produces similar results to the laser device (red LASER 635nm) when preformed using a specified treatment protocol.

Furthermore, it is hypothesized that the Vevazz therapy program achieves the results after one 28 minute treatment period. The predicate 635nm LED device (Photonica Professional by Ward Photonics) achieves its results after one 32 minute therapy program.

The FB Professional therapy program uses the FB Professional LED device for fat removal using LED red light therapy. This multi-site study reviews results from 70 randomly selected patients after a single treatment using the FB Professional LED device.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older.
* May be male or female.
* Generally good health.

Exclusion Criteria:

* Minors.
* Open wounds or sores.
* Pacemaker.
* Photosensitivity.
* Epilepsy.
* Any form of cancer.
* Severe kidney or liver problems.
* Thyroid problems.
* Pregnant or nursing.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fat Amount (Reduction) in Treatment Area as Measured in Inches Lost | One 28 minute session
  Circumferential measurement of thighs, hips and waist before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ligertwood, Dr, Principal Investigator — Human Studies Group
Locations (1):
- Ligertwood Chiropractic, New Port Richey, Florida, United States